CLINICAL TRIAL: NCT02483221
Title: Phase 4 Study of Postoperative Pain Therapy With Hydromorphone Using Patient-Controlled Target-Controlled Infusion (TCI-PCA) vs. Patient-Controlled Analgesia (PCA) With Morphine After Elective Cardiac Surgery
Brief Title: Postoperative Pain Therapy With Hydromorphone TCI-PCA vs. Morphine PCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCI-PCA-002
Record Dates: First submitted 2015-06-24; First posted 2015-06-26 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Acute Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Hydromorphone; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCI-PCA (Active Comparator)
  Interventions: Drug: Hydromorphone
- PCA (Active Comparator)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Hydromorphone — Hydromorphone is given intravenously by TCI-PCA. The TCI-PCA system steer the hydromorphone infusion pump to achieve plasma and effect-site concentrations of hydromorphone in predefined increasing steps on patient request and in predefined decreasing steps on lack of patient request within predefined plasma and effect-site concentration range, lockout times and infusion speed.
  Arms: TCI-PCA
Drug: Morphine — Morphine is given intravenously by PCA. The PCA pump administers a predefined bolus dose on patient request considering the predefined lockout time and infusion speed.
  Arms: PCA

SUMMARY:
Treatment of postoperative pain with hydromorphone (a strong analgesic) using patient-controlled analgesia with target-controlled infusion compared to conventional patient-controlled analgesia with morphine after elective cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Scheduled for elective cardiac surgery involving thoracotomy and subsequent ICU stay

Exclusion Criteria:

* Administration of other analgesics or sedatives, if not administered in stable dosages for at least 14 days or if not used for premedication and surgery
* Administration of hydromorphone or morphine in the period between screening and surgery
* Severe hepatic or renal impairment in medical history
* BMI>= 35 ASA>= 4

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Score | up to 17 hours after extubation
  Comparison of pain analgetic efficacy between hydromorphone TCI-PCA and conventional morphine PCA during the early postoperative stage

SECONDARY OUTCOMES:
Modified Observer's Assessment of Alertness/Sedation Scale | up to 17 hours after extubation
  Comparison of opioid induced sedation level between hydromorphone TCI-PCA and conventional morphine PCA during the early postoperative stage
Postoperative Nausea and Vomiting | day of surgery
  Comparison of opioid associated nausea and vomiting between hydromorphone TCI-PCA and conventional morphine PCA during the early postoperative stage
Respiratory Frequency | up to 17 hours after extubation
  Comparison of opioid induced respiratory depression between hydromorphone TCI-PCA and conventional morphine PCA during the early postoperative stage

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jeleazcov, MD, MS, Principal Investigator — Department of Anesthesiology, University Hospital Erlangen
Locations (1):
- Department of Anesthesiology, University Hospital Erlangen, Erlangen, Bavaria, Germany

REFERENCES:
- [Derived] Ihmsen H, Schuttler J, Jeleazcov C. Pharmacokinetics of Morphine and Morphine-6-Glucuronide During Postoperative Pain Therapy in Cardiac Surgery Patients. Eur J Drug Metab Pharmacokinet. 2021 Mar;46(2):249-263. doi: 10.1007/s13318-020-00663-z. Epub 2021 Feb 5. PMID 33547559